CLINICAL TRIAL: NCT05977647
Title: Comparison of Silodosin Versus Tamsulosin on Passage of Acutely Obstructing Ureteral Calculi (History of Last 4 Weeks) in Medical Expulsive Therapy
Brief Title: Medical Stone Expulsive Therapy for Acutely Obstructed Ureteric Calculi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-MSE-001-23
Record Dates: First submitted 2023-07-07; First posted 2023-08-04 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Ureteric Stone of Lower Third of Ureter
MeSH Terms: interventions — Tamsulosin; silodosin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups.
  1. A permuted block randomization technique will be used
  2. A block represents a separate center/site of enrollment.
  3. There will be 19 recruitment centers
  4. Each center will enroll total 20-25 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Active Comparator): Patients with lower ureteric stone will be randomized through permuted block randomization equally into two group. 120 patients will be on tamsulosin 0.4 mg once daily, therapy will be given for a maximum of 4 weeks.
  Interventions: Drug: Tamsulosin Oral Capsule
- Silodosin (Active Comparator): Patients with lower ureteric stone will be randomized through permuted block randomization equally into two group. 120 patients will be on Silodosin 8 mg once daily. Therapy will be given for a maximum of 4 weeks.
  Interventions: Drug: Tamsulosin Oral Capsule

INTERVENTIONS:
Drug: Tamsulosin Oral Capsule — Patient will be enrolled in one of study arm through randomization.
  Other Names: silodosin Oral Capsule

SUMMARY:
As a first treatment option for small-size ureteric stones, α-blockers are now being used for medical expulsive therapy (MET) instead of invasive procedures. There is high evidence of the therapeutic benefit of α-blockers in the treatment of Distal ureteric stone (DUS); also endorsed by international guidelines.

However, limited data is available worldwide, on the effect of silodosin to treat DUS. A multi-center study is needed to confirm the efficacy and safety of therapy.

DETAILED DESCRIPTION:
A kidney stone is a crystal formed inside the kidney. It is one of the commonest conditions of kidney disease affecting 12% of the world's population. Out of 12% Ureteric stones, around 20% represent cases of urolithiasis, of which 70% are situated in the lower third of the ureter and are termed as 'Distal Ureteric Stones' (DUS). Kidney stone aggravates the risk of end-stage kidney disease and increases the risk of multiple complications. including chronic kidney disease hypertension, diabetes, and cardiovascular diseases. The commonest type of kidney stone is calcium oxalate, which is present in around 70 to 80% of the total reported cases of kidney stones.

There are multiple approaches to the management of ureteric stones, which has evolved over the last 20 years, specifically due to advancements in technology, use of ureteroscopy and shockwave lithotripsy (SWL) as minimally invasive treatment options. However, these interventions are quite expensive and may lead to multiple complications. According to the complication rate of minimally invasive interventions is 2.5%.

As a first treatment option for small-size ureteric stones, α-blockers are now being used for medical expulsive therapy (MET) instead of invasive procedures. As observed through two meta-analyses there is high evidence of the therapeutic benefit of α-blockers in the treatment of DUS seen to be 52% and 44% higher than those patients who have not received any treatment.

There is an endorsement of the use of a-blockers as a management option for ureteric stones by the American Urology Association (AUA) and the European Association of Urology. The α1A- adrenoceptors have proven to play an important effect in intervening contraction of the human ureter, induced by phenylephrine. Silodosin (selective α1-adrenoceptor blocker) in the human ureter was found more efficacious than Tamsulosin (1D-adrenoceptor blocker) in non-adrenaline-induced contractions.

However, limited data is available worldwide, on the effect of silodosin to treat DUS. To the best of our knowledge, there has been no study done on the use of silodosin as MET for DUS in the context of Pakistan. Therefore, this study will be able to provide meaningful data to find the efficacy and safety of silodosin in comparison to Tamsulosin as MET in ureteric stone.

ELIGIBILITY:
Inclusion Criteria:

* Adults male and female aged 18 to 70 years
* Patients who give informed consent
* Stone located in the distal 1/3rd of ureter (Single, unilateral and radiopaque ureteral calculus 5 to 10 mm visible on the CT-KUB± X-ray KUB within the ureter
* Serum creatinine level within the normal range (adult men, 0.74 to 1.35 mg/dL & 0.59 to 1.04 mg/dL)
* Ability to tolerate oral fluids and oral pain medication

Exclusion Criteria:

* Patients already taking an alpha-adrenergic antagonist medication for 4 weeks
* Evidence of any other renal stone simultaneously present or at any location
* Hydronephrosis Grade 3 (Moderate) & Grade 4 (Severe) Patients with eGFR <60 ml/min/1.73m2
* Signs of infection including temperature >38ºC or Urinalysis with any of the following: Positive Leukocyte Esterase, Positive Nitrates, or White Blood Cell Count >5/hfp in the setting of a positive urine culture (defined as a single isolated bacterial species population of >100,000 CFU)
* Patients with chronic pain already undergoing treatment with narcotic medications or drug abusers
* Pregnant or lactating women
* Patient suffering from urinary tract infection, ureteral surgery, and existing DJ stents.
* Clinical jaundice
* Any forms of anatomical obstructions in the urinary tract
* The previously suffering from postural hypotension
* Any other disease jeopardizing participation in trial and could lead to increase patient health risks
* History of allergic reactions with the study drugs (Silodosin or Tamsulosin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
% of stone expulsion | 4 weeks
  The primary outcome measure will be the passage of stone expulsion self-reported definitive passage of calculus or the first day of pain-free to 48 hours period with calculus absent of X - ray KUB.

SECONDARY OUTCOMES:
Time in days to stone expulsion | 4 weeks
  Time in days to stone expulsion: Self-reported definitive passage of calculus or the first day of pain-free to 48 hours period with calculus absent of X - ray.
Frequency of pain reported by patients | 4 weeks
  Patient will mark the number of episodes of pain in 24 hours on daily basis in patient dairy..
Change in intensity of pain | 4 weeks
  Patient dairy will be provided to all the patients. Which will have pain log scale. They will self-report the intensity of pain (highest intensity) in 24 hours on daily basis. The pain scale ranges are mentioned below.
  1. 0 means no pain
  2. 1 to 2 means mild pain
  3. 2 to 4 means moderate pain
  4. 4 to 6 means severe pain
  5. 6 to 8 means very severe pain
  6. 8 to 10 means worst pain ever
Usage of analgesics | 4 weeks
  The subject will be given a standardized pain medication (diclofenac sodium) prescription at their initial visit and will be asked to keep track of how much pain medication they used each day in patient's dairy. This information will be collected at every week on follow up visits.
Frequency of ER visits | 4 weeks
  Patient will report if he/she had visited ER in last 24 hours on daily basis in patient's dairy along with the medication prescribed in ER.
Frequency of adverse events (Postural hypotension, retrograde ejaculation, etc.) | 4 weeks
  Patient will be briefed about the known adverse events of study drugs. If any side effects is observed by the patient will be reported in patient dairy.
  If any unknown side effects happen that will also be reported in patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Salman El Khalid, MBBS, Principal Investigator — The Kidney Centre
Locations (1):
- North west general hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No